CLINICAL TRIAL: NCT05503173
Title: Integrated Telehealth Intervention To Reduce Chronic Pain And Unhealthy Drinking Among People Living With HIV (PLWH)
Brief Title: Telehealth for Pain and Unhealthy Drinking Among PLWH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-42405; 1P01AA029546-01 (NIH)
Record Dates: First submitted 2022-08-13; First posted 2022-08-16 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: HIV; Chronic Pain; Unhealthy Alcohol Use
Keywords: Pain management; Telehealth; Unhealthy drinking; Ecological momentary assessment
MeSH Terms: conditions — Chronic Pain; Agnosia | interventions — Crisis Intervention; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational and Cognitive-Behavioral Management for Alcohol and Pain Intervention (MCBMAP) (Experimental): Participants randomized to this arm will receive MCBMAP which utilizes a self-regulation framework to integrate evidence-based approaches for chronic pain and unhealthy drinking.
  Interventions: Behavioral: MCBMAP
- Brief Advice and Information (Active Comparator): Participants randomized to this arm will be provided treatment as usual for their conditions.
  Interventions: Other: Brief Advice and Information

INTERVENTIONS:
Behavioral: MCBMAP — MCBMAP integrates motivational interviewing (MI) and cognitive-behavioral skill training interventions for unhealthy drinking with cognitive-behavioral and self- management approaches for chronic pain. The intervention is delivered through internet-based videoconferencing and supplemented with web-based content to support the intervention. The initial treatment session provides a rationale for addressing alcohol and pain together in the context of HIV management, and initiates MI related to alcohol use. Participants receive 6 additional treatment sessions over the subsequent weeks.
  Arms: Motivational and Cognitive-Behavioral Management for Alcohol and Pain Intervention (MCBMAP)
Other: Brief Advice and Information — Through videoconferencing an interventionist will provide participants psychoeducation about the effects of alcohol and pain on HIV symptoms, advice/recommendations to reduce alcohol use, and a list of local treatment resources for alcohol and chronic pain.
  Other Names: Treatment as usual
  Arms: Brief Advice and Information

SUMMARY:
This randomized controlled trial is a between-groups design to compare the Motivational and Cognitive Behavioral Management for Alcohol and Pain (MCBMAP) Intervention to a Brief Advice and Information Control condition.

Two-hundred and fifty participants who have HIV with moderate or greater chronic pain will be randomized for the trial. Recruitment will take place through digital media. A unique feature of this intervention trial is that most of the procedures will be conducted remotely which will minimize barriers of transportation and time for participants. Consent and baseline assessment will be completed remotely. Following baseline assessment, participants will complete two weeks of ecological momentary assessment (EMA) to assess alcohol use, chronic pain, physical function and mechanisms of behavior change for alcohol and pain management. Following the two-week phase, participants will be randomly assigned to either the intervention or control condition and meet the interventionist through videoconferencing. Participants will complete outcome assessment measures at 3- and 6-months post-baseline. Following the 3-month outcome assessment, participants will complete another two weeks of EMA.

ELIGIBILITY:
Inclusion Criteria:

* Able to confirm HIV diagnosis, via visual evidence of antiretroviral (ART) medication bottle or medical record presented to study staff over Zoom.
* Engaged in unhealthy drinking, defined as:
* >7 drinks for women / > 14 drinks for men per week.
* OR ≥ 3 drinks for women / ≥4 drinks for men on one occasion in the past month.
* Experiencing moderate or greater chronic pain (4 or greater on the numerical pain rating scale) for at least 3 months.
* Own a smart phone.
* Lives in the USA.
* Has a US mailing address.

Exclusion Criteria:

* History of bipolar, schizoaffective disorder or schizophrenia per self report.
* Unstable dose of psychoactive medication for pain or alcohol/substance use [i.e., if on medication, participant has not been on same dose for least 2 months]
* History of withdrawal-related seizures or delirium tremens
* Current non-pharmacological treatment for alcohol use disorder or chronic pain
* Acute life-threatening illness that requires treatment or intend to have surgery for a pain-related condition in the next 6-months.
* Current cancer-related pain
* Unable to provide one or more individuals for follow-up contact
* Individual who is unwilling to provide their sex at birth
* Limited or non-readers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of alcoholic drinks consumed per week at 6 months | 6 months
  Assessed by the Timeline Follow Back (TLFB-30) which is a is a calendar that allows an assessor to obtain an estimate of an individual's daily drinking habits over a 30-day time period.
Number of heavy episodic drinking days the past month at 6 months | 6 months
  Assessed by the Timeline Follow Back (TLFB-30) which is a is a calendar that allows an assessor to obtain an estimate of an individual's daily drinking habits over a 30-day time period.
Rating of pain severity and interference at 6 months | 6 months
  Assessed by the PEG Scale Assessing Pain Intensity and Interference (PEG) which is a 3-item scale measuring pain intensity, emotional function, and physical function over the past week.

SECONDARY OUTCOMES:
Rating of pain severity at 6 months | 6 months
  Assessed by the Brief Pain Inventory (BPI) which a 9-item self-report questionnaire in which participants rate the severity of pain and the degree of pain interference with various dimensions of feeling and function. Related pain is rated on a 0-10 scale and scored as Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Rating of pain interference at 6 months | 6 months
  Assessed by the Brief Pain Inventory (BPI) which a 9-item self-report questionnaire in which participants rate the severity of pain and the degree of pain interference with various dimensions of feeling and function. Related pain is rated on a 0-10 scale and scored as Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tibor P Palfai, PhD, Principal Investigator — Boston Medical Center, Psychiatry; BU Psychological & Brain Sciences
Locations (1):
- Charles River Campus, Boston University, Psychology Department- remote study, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palfai TP, Bernier LB, Kratzer MP, Magane KM, Fielman S, Otis JD, Heeren TC, Winter MR, Stein MD. Integrated telehealth intervention to reduce chronic pain and unhealthy drinking among people living with HIV: protocol for a randomized controlled trial. Addict Sci Clin Pract. 2024 Sep 5;19(1):64. doi: 10.1186/s13722-024-00493-3. PMID 39238059